CLINICAL TRIAL: NCT06335927
Title: Hepatic Arterial Infusion Chemotherapy Combined With Cadonilimab and Regorafenib as Second-line Treatment for Unresectable Intrahepatic Cholangiocarcinoma: a Single-arm, Phase II Study
Brief Title: HAIC Combined With Cadonilimab and Regorafenib as 2nd-line Treatment for ICC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Director of Hepatobiliary Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWK2023-001
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: HAIC; Cadonilimab; Regorafenib; Second-line; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAIC-GEMOX+Cadonilimab+Regorafenib (Experimental): HAIC-GEMOX: Gemcitabine 1000mg/m2 on Day 1 + Oxaliplatin 85mg/m2 on Day 1, every 3 weeks (Q3W), for up to 6 treatment cycles in combination with Cadonilimab (6mg/kg, D2, Q3W) and Regorafenib (80mg QD, Q3W)
  Interventions: Drug: HAIC-GEMOX+Cadonilimab+Regorafenib

INTERVENTIONS:
Drug: HAIC-GEMOX+Cadonilimab+Regorafenib — HAIC-GEMOX: Gemcitabine 1000mg/m2 on Day 1 + Oxaliplatin 85mg/m2 on Day 1, every 3 weeks (Q3W), for up to 6 treatment cycles in combination with Cadonilimab (6mg/kg, D2, Q3W) and Regorafenib (80mg QD, Q3W)

SUMMARY:
This study is a single-arm Phase II clinical trial aiming to evaluate the safety and efficacy of HAIC combined with Cadonilimab and Regorafenib as second-line treatment for unresectable intrahepatic cholangiocarcinoma.

The study plans to enroll approximately 45 participants. All enrolled participants will receive continuous treatment: HAIC-Gemox: Gemcitabine 1000mg/m2 on Day 1 + Oxaliplatin 85mg/m2 on Day 1, every 3 weeks (Q3W), for up to 6 treatment cycles, Cadonilimab(6mg/kg, D2, Q3W) and Regorafenib (80mg QD, Q3W) until the investigator determines that there is no longer any clinical benefit (based on comprehensive assessment including RECIST v1.1 imaging evaluation and clinical condition), intolerable toxicity, initiation of new anti-tumor therapy, or meeting other criteria for treatment discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment in the study, participants must meet the following inclusion criteria:

1. Voluntarily provide written informed consent.
2. Age at enrollment is ≥18 years and ≤75 years, both males and females.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Expected survival period of ≥3 months.
5. Patients with histologically or cytologically confirmed unresectable intrahepatic cholangiocarcinoma. Patients who have failed standard treatment (standard treatment includes gemcitabine plus cisplatin plus pembrolizumab, gemcitabine plus gemcitabine plus oxaliplatin, capecitabine plus oxaliplatin, chemotherapy mainly based on albumin-bound paclitaxel, 5-fluorouracil (5-FU) plus platinum-based therapy) or are intolerant to standard treatment, or patients for whom standard treatment is not accessible. Note: Patients who have received adjuvant/neoadjuvant chemotherapy targeting non-metastatic disease with curative intent and experience disease progression within ≤6 months after the last treatment are eligible.
6. At least one measurable lesion according to RECIST v1.1 that can be accurately measured repeatedly. Note: Brain metastases cannot be considered as target lesions.
7. Adequate organ function determined by the following requirements:

   1. Hematology (no use of any blood components or growth factors within 7 days prior to starting the study treatment): i. Absolute Neutrophil Count (ANC) ≥ 1.5 × 109/L (1,500/mm3). ii. Platelet count ≥ 80 × 109/L (100,000/mm3). iii. Hemoglobin ≥ 90 g/L.
   2. Kidney:

   i. Serum creatinine ≤ 1.5 × Upper Limit of Normal (ULN). ii. Calculated creatinine clearance* (CrCl) ≥ 50 mL/min.

   * CrCl will be calculated using the Cockcroft-Gault formula (Cockcroft-Gault formula).

   CrCl (mL/min) = {(140 - age) × body weight (kg) × F} / (SCr (mg/dL) × 72) For males, F = 1; for females, F = 0.85; SCr = serum creatinine. iii. Urine protein ≤ 1+ or 24-hour urinary protein quantification < 1.0 g. c) Liver: i. Total bilirubin (TBil) ≤ 3 × ULN. ii. AST and ALT ≤ 5 × ULN. iii. Serum albumin (ALB) ≥ 28 g/L. d) Coagulation function: i. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN (unless the subject is receiving anticoagulant therapy and coagulation parameters [PT/INR and APTT] are within the expected range for anticoagulant treatment at screening).

   e) Cardiac function: i. Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
8. Female participants of childbearing potential must undergo urine or serum pregnancy testing within 3 days prior to the first dose of study medication (if the urine pregnancy test results cannot be confirmed as negative, a serum pregnancy test must be conducted, with the serum pregnancy test result being definitive). If female participants of childbearing potential engage in sexual activity with a nonsterilized male partner, they must use an acceptablemethod of contraception from the start of screening and agree to continue using contraception for up to 120 days after the last dose of the study medication. The decision to stop contraception after this time should be discussed with the investigator.
9. Male participants with a female partner of childbearing potential must use effective contraception from the start of screening until 120 days after the last dose of the study medication. The decision to stop contraception after this time should be discussed with the investigator.
10. Participants must be willing and able to comply with the scheduled visits, treatment plan, laboratory tests, and other study requirements.

Exclusion Criteria:

Subjects meeting any of the following criteria will be ineligible to participate in this study:

1. Diagnosis of malignant tumors with non-biliary cancers such as hepatocellular carcinoma, mixed-cell carcinoma, or fibrolamellar carcinoma.
2. History of other malignant tumors within the past 3 years, except for cured localized tumors (e.g., basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ).
3. Concurrent participation in another clinical study unless it is an observational, non-interventional study or follow-up period of an interventional study.
4. Palliative local therapy performed on non-target lesions within 2 weeks prior to the first dose; non-specific immune modulating therapy (e.g., interleukins, interferons, thymosin, excluding IL-11 for thrombocytopenia) within 2 weeks prior to the first dose; use of traditional Chinese medicine or herbal remedies with anti-tumor indications within 1 week prior to the first dose.
5. Previous receipt of any immune anti-tumor therapy, including immune checkpoint stimulants (e.g., ICOS, CD40, CD137, GITR, OX40 antibodies), immune cell therapy.
6. Previous receipt of targeted therapy.
7. Active autoimmune diseases requiring systemic treatment within the past two years (e.g., medications for disease improvement, corticosteroids, immunosuppressive therapy); replacement therapy (e.g., thyroid hormones, insulin, physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic treatment.
8. History of active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea).
9. History of immunodeficiency; positive HIV antibody test; current long-term use of systemic corticosteroids or other immunosuppressive agents.
10. Known active tuberculosis (TB) or suspected active TB requiring clinical evaluation; known active syphilis infection.
11. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
12. History of or current non-infectious pneumonitis/interstitial lung disease requiring systemic corticosteroid therapy.
13. Severe infection within 4 weeks prior to the first dose, including complications requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective treatment within 2 weeks prior to the first dose (excluding antiviral therapy for hepatitis B or C).
14. Subjects with active hepatitis B (positive HBsAg and HBV-DNA >1000 copies/mL [200 IU/mL] or above the lower limit of detection, whichever is higher). Note: Subjects with hepatitis B should receive antiviral therapy during the study treatment period.
15. Subjects with active hepatitis C (positive HCV antibody and HCV-RNA above the lower limit of detection).
16. Presence of obstructive jaundice (eligible if actively treated with biliary drainage or stenting and liver function has recovered).

    Major surgery or significant traumatic injury within 30 days prior to the first dose, or planned major surgery within 30 days after the first dose (as determined by the investigator); minor surgical procedures within 3 days prior to the first dose (excluding placement of peripheral intravenous catheters and implantation of venous infusion ports).
17. Subjects with active central nervous system (CNS) metastases. Note: Subjects with previously treated brain metastases (e.g., surgery, radiotherapy) may be eligible if clinically stable for at least two weeks after treatment (from the start of study drug administration) and off corticosteroids for three days prior to study drug administration. Subjects with untreated, asymptomatic brain metastases (i.e., no neurological symptoms, no requirement for corticosteroids, and no brain metastases with a longest diameter >1.5 cm) may be eligible and should have regular assessments of brain metastases during the course of the study treatment.
18. Known brainstem, meningeal, spinal cord, or leptomeningeal metastases or compression.

    Subjects with clinically significant symptoms or requiring repeated drainage of pleural effusion, pericardial effusion, or ascites.

    Inability to swallow tablets, malabsorption syndrome, or any condition that could affect gastrointestinal absorption.
19. Current uncontrolled concurrent illness, including but not limited to decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorder, severe active peptic ulcer disease or gastritis, or any psychiatric/social condition that would limit compliance with study requirements or affect the subject's ability to provide written informed consent.
20. History of myocarditis, cardiomyopathy, malignant arrhythmia. Subjects with unstable angina, myocardial infarction, congestive heart failure (New York Heart Association functional class II or higher), or vascular disease with a risk of rupture requiring hospitalization within 12 months prior to the first dose of study drug, or other cardiac damage (e.g., poorly controlled arrhythmias, myocardial ischemia) that may affect the assessment of the safety of the study drug.
21. History within 6 months prior to the first dose of study drug of esophageal or gastric variceal bleeding, severe ulceration, unhealed wound, gastrointestinal perforation, fistula, intra-abdominal abscess, or acute gastrointestinal bleeding; any arterial thromboembolic event within 6 months prior to the first dose of study drug, grade 3 or higher venous thromboembolism according to NCI CTCAE version 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy; current hypertension with a systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg after oral antihypertensive therapy.
22. History of severe bleeding diathesis or coagulation disorder; clinically significant bleeding symptoms within 1 month prior to the first dose of study drug, including but not limited to gastrointestinal bleeding, bleeding gastric ulcer, hemoptysis (defined as coughing or spitting up ≥1 teaspoon of fresh blood or small clots or coughing blood without sputum, subjects with blood-tinged sputum are allowed), epistaxis (excluding nosebleeds and regurgitant epistaxis); subjects receiving continuous anticoagulant therapy within 10 days prior to the first dose of study drug.
23. Screening imaging showing tumor encasement or invasion of major blood vessels or organs (such as heart and pericardium, trachea, esophagus, aorta, superior vena cava, etc.) or presence of significant necrosis, cavitation, and the investigator determines that entry into the study would pose a risk of bleeding.
24. Previous unresolved toxicity from anticancer treatment, defined as toxicity not recovered to grade 0 or 1 according to NCI CTCAE version 5.0 or as specified in the inclusion/exclusion criteria, except for alopecia and residual neurotoxicity related to previous platinum-based treatment. Subjects with irreversible toxicity that is not expected to worsen with study drug administration (e.g., hearing loss) may be considered for inclusion in the study after consultation with the investigator. Subjects with late toxicities caused by radiotherapy that the investigator deems irrecoverable may be considered for inclusion in the study.
25. Administration of live vaccines within 30 days prior to the first dose or planned administration of live vaccines during the study is not allowed, but the use of inactivated vaccines is permitted.
26. Known allergies to any component of the investigational drug or a history of severe hypersensitivity reactions to other monoclonal antibodies.
27. Known history of mental illness, substance abuse, alcoholism, or drug addiction.
28. Pregnant or lactating women.
29. Previous or current presence of any condition, treatment, or laboratory abnormalities that may confound study results, affect the subject's full participation in the study, or be contrary to the subject's best interests.
30. Non-malignant diseases causing local or systemic symptoms or conditions secondary to the tumor, leading to higher medical risks and/or uncertainty in survival assessment, such as tumor-related leukemic reaction (white blood cell count >20 × 109/L), manifestations of cachexia (e.g., known weight loss exceeding 10% in the 3 months before screening), etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 54 weeks
  Objective Response Rate (ORR), based on RECIST v1.1 assessment.

SECONDARY OUTCOMES:
Hepatic Objective Response Rate (hORR) | 54 weeks
  Hepatic Objective Response Rate (hORR) based on RECIST v1.1 assessment.
Duration of Response (DoR) | 54 weeks
  Duration of Response (DoR) based on RECIST v1.1 assessment.
Disease Control Rate (DCR) | 54 weeks
  Disease Control Rate (DCR) based on RECIST v1.1 assessment.
Time to Response (TTR) | 54 weeks
  Time to Response (TTR) based on RECIST v1.1 assessment.
Progression-Free Survival (PFS) | 54 weeks
  Progression-Free Survival (PFS)
Overall Survival (OS) | Up to approximately 5 years
  Time from enrollment to death
Safety and tolerability | 54 weeks
  Incidence of Adverse Events and Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China